CLINICAL TRIAL: NCT02491645
Title: Comparison of Effectiveness of Home Based Sensory Interventions Along With Standard Therapy Versus Standard Therapy Alone in Autistic Children With Sensory Processing Abnormalities :An Open Label Randomized Study
Brief Title: Comparison of Effectiveness of Home Based Sensory Interventions Along With Standard Therapy Versus Standard Therapy Alone in Autistic Children With Sensory Processing Abnormalities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr Hansashree P, Senior resident , pursuing DM Pediatric neurology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PGIMER-HS
Record Dates: First submitted 2015-07-03; First posted 2015-07-08 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Autistic Children With Sensory Processing Abnormalities
Keywords: Autistic spectrum disorder; Sensory processing abnormalities; Sensory interventions; occupational therapy
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Children would receive both standard therapy and home based sensory interventions as described below,
  * Standard therapy - children would receive measures like speech and language services, behavioral interventions and educational program regularly as and when decided by the primary care physician. They would be individualized to child specific needs .
  * Home based sensory interventions - children would receive home based sensory interventions targeting visual and auditory system, tactile abnormalities, proprioceptive and vestibular abnormalities.These interventions would be carried out daily , at least 5 days a week, for a minimum duration of 1hour/day.
  Interventions: Other: Sensory interventions
- Control group (No Intervention): This group of children would receive only standard therapy as described below, Standard therapy - children would receive measures like speech and language services, behavioral interventions and educational program regularly as and when decided by the primary care physician. They would be individualized to child specific needs.

INTERVENTIONS:
Other: Sensory interventions — 1. Tactile stimulation: Brushing technique , handling materials of various textures, bear hug and rug , play dough and find in rice techniques to be done.
  2. Proprioception technique : Joint compression , popping bubbles, lifting weights of different measures and scooter board push activities to be done.
  3. Movement/vestibular techniques :Bear hug and rug , swinging or rocking motion, jumping or spinning to be done.
  4. Visual stimulation : picture recognition, dot colouring , lighting balls and toys , familiarisation of emotions to be done.
  5. Auditory stimulation : Sound familiarisation and music time will be done.
  Arms: Intervention group

SUMMARY:
Around 69-95% of children with Autistic Spectrum Disorder are known to have sensory processing abnormalities .Tackling these problems would help in better quality of life, both for the parents and the children. Sensory integration therapy, an individualized clinic based therapy have been shown to have a positive effect on those children with sensory abnormalities. Hence the investigators are doing this study , to primarily look into the efficacy and feasibility of home based sensory interventions in autistic children with sensory processing abnormalities.

ELIGIBILITY:
Inclusion Criteria:

1. Children between the age group of 3-12years with autistic spectrum disorder as per DSM -V criteria along with CARS and those having sensory abnormalities as screened by short sensory profile 2 will be included in the study group
2. Parents who agreed for home based sensory intervention therapy with strict adherence to same and to refrain from initiation of any new treatments including medications during study period

Exclusion Criteria:

1. Children with epileptic syndromes with language regression(LKS)
2. Children with features of ASD but having underlying structural(TS), neurometabolic or primary epilepsy as etiology
3. Children with uncontrolled seizures (seizures in the last 06 months)
4. Children whose parents do not give consent for the study
5. Children for whom follow up would not be feasible

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2015-02; Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
1. Comparison of change in total score on 10 item Likert scale (as rated by parents) | 3 months

SECONDARY OUTCOMES:
1. Comparison of change in health related quality of life using PedsQL ( Pediatric quality of life inventory) questionnaire | 3 months
2. Comparison of change in overall functional outcome using CGAS (Children's global assessment scale) questionnaire | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Hansashree Padmanabha, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Dr Hansashree P, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No